CLINICAL TRIAL: NCT05959642
Title: Comparing Controlled Flow Delivery Dentapen® Technique to Traditional Syringes on Pain Perception During the Administration of Anesthesia Among A Group of Pediatric Dental Patients: A Split-Mouth Randomized Clinical Trial
Brief Title: Comparing Controlled Flow Delivery Dentapen® Technique to Traditional Syringes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, reham salman alshakhs, Master Degree Student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Denta pen
Record Dates: First submitted 2023-05-17; First posted 2023-07-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Early Childhood Caries
Keywords: non invasive technique

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled Flow Delivery Dentapen (Experimental): Controlled Flow Delivery Dentapen - infiltration upper d according to the manufacturer instructions it works with standardised 1.8 ml local anaesthetic carpules . 1)we raise the lip a little 2) we use dentapen for anaesthesia 3) class 1 cavity preparation Articaine hydrochloride 4% with 1:100,000 epinephrine will be injected.The dentist will wait 5 seconds
  Interventions: Device: dentapen
- Traditional metal Syringes (Active Comparator): Traditional metal Syringes we raise the lip a little 2) infiltration upper d we use traditional syringes 3)class 1 cavity preparation with composit filling works with standardised 1.8 ml local anaesthetic carpules . we use Articaine hydrochloride 4% with 1:100,000 epinephrine will be injected.The dentist will wait 5 seconds
  Interventions: Device: Traditional metal Syringes

INTERVENTIONS:
Device: dentapen — Experimental: Controlled Flow Delivery Dentapen according to the manufacturer instructions, It works with standardised 1.8 mL local anaesthetic carpules. The distalingual and mesiolingual line angles are the most effective for multi-rooted upper D teeth.
  Articaine hydrochloride 4% with 1:100,000 epinephrine will be injected for each root as shown on a special indicator.The dentist will wait 5 seconds before needle withdrawal. Same steps will be repeated at the mesiolingual line angle
  Arms: Controlled Flow Delivery Dentapen
Device: Traditional metal Syringes — Active Comparator: Conventional Injection of infiltration upper d a standard technique for the Injection of infiltration upper d will be used supplemented with long buccal infiltration for the buccal gingiva.
  A 27-gauge disposable dental needle will be used to inject Articaine hydrochloride 4% with 1:100,000 epinephrine. The needle will be directed to primary molars
  Arms: Traditional metal Syringes

SUMMARY:
This study compares the effect of the controlled flow delivery Dentapen® technique to traditional syringes on pain perception during dental procedures among a group of pediatric dental patients

DETAILED DESCRIPTION:
Local anesthetic injections are usually the main reason for fear and anxiety during dental treatment. Pain management is a critical aspect of pediatric dental care. Fear associated with seeing and experiencing needle penetration, sensation of swelling soft tissues and prolonged numbness as well as allergic reactions to the anesthetic fluid, are the most common factors causing patients and dental clinicians to experience anxiety regarding the use of infiltration local anesthesia. Exploring new alternative and a traumatic method will help improving the quality of care in pediatric dentistry.

Consequently, there is a constant search for new techniques looking to avoid the invasive and often painful nature of the anaesthetic injection required for dental treatments, making it a more pleasant and less distressing experience for patients.

Even though there are no techniques available that can totally replace conventional local anaesthesia, some alternatives have been developed that are effective in a limited range of procedures. In 1997, a new method for the administration of anaesthetics was launched: the computer- controlled local anaesthesia delivery system (CCLADS). After

2006, the single tooth anaesthesia system (STA) (Milestone Scientific, Inc. Livingston, NJ, USA) was also introduced.

Currently, one of the most discouraging aspects for many patients undergoing dental procedures is the administration of anaesthesia. Consequently, there is a constant search for new techniques to avoid the invasive and painful nature of the injection. A new, cableless, motorised syringe system (Dentapen®) has recently been developed, standing out for its convenience and ease of use. The slow injection of anaesthetics at low pressure appears to reduce pain and discomfort during dental anaesthesia, and that currently does not require specific training. It has several injection settings, allowing it to be held like a syringe or pen, and is compatible with all anaesthetic needles and cartridges from all brands with an accurate control of flow and pressure of the injection can therefore mitigate the pain experienced by these patients.

So, the purpose of the current study was to evaluate the effect of controlled flow delivery Dentapen® technique on pain perception among a group of pediatric dental patients in comparison to conventional injection technique.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6 and 8 years

  * Healthy children with no systemic problems.
  * Cooperative Children
  * First dental visit
  * Children willing to provide assent and parent willing to provide informed consent
  * Bilaterally decayed primary maxillary first molars with normal radiographic findings and need restorative treatment

Exclusion Criteria:

Children with previously restored teeth

* Children requiring emergency dental treatment (cellulitis, abscess)
* Children's teeth with signs or symptoms of Pulpitis
* Children whose parents refuse to sign the informed consent.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain perception during injection of local anesthesia | in the same visit after finishing the procedure, 0 scale - no pain , 10 scale -worest
  Wong-Baker faces pain rating scale; Scores (0-10)

SECONDARY OUTCOMES:
Heart rate during injection of local anesthesia | in the same visit after finishing the procedure
  measured by Pulse oximeter, Beats per minute (BPM)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carvajal-Nunez U, Prieur D, Vitova T, Somers J. Charge distribution and local structure of americium-bearing thorium oxide solid solutions. Inorg Chem. 2012 Nov 5;51(21):11762-8. doi: 10.1021/ic301709d. Epub 2012 Oct 16. PMID 23072315